CLINICAL TRIAL: NCT03428633
Title: Thoracic Paravertebral Blocks in Open Nephrectomy. A Prospective, Randomized Study of Block Efficacy and Influence on Oxidative Stress and Patient Outcome.
Brief Title: Thoracic Paravertebral Blocks in Open Nephrectomy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Asklepieion Voulas General Hospital (Other Government)
Collaborators: Michail Tsagkaris (Unknown); Chryssoula Staikou (Unknown); Ioannis Karavokyros (Unknown)
Responsible Party: Principal Investigator, Alexandros Makris, Consultant Anaesthesiologist, Asklepieion Voulas General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AsklepieionVGH
Record Dates: First submitted 2018-02-01; First posted 2018-02-09 (Actual); Last update posted 2023-10-13 (Actual); Status verified 2023-10

CONDITIONS: Nephrectomy; Analgesia
MeSH Terms: conditions — Agnosia | interventions — Ropivacaine; Morphine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator): Thoracic paravertebral block using ropivacaine
  Interventions: Drug: Ropivacaine
- Group B (Active Comparator): Morphine IV
  Interventions: Drug: Morphine

INTERVENTIONS:
Drug: Ropivacaine — Paravertebral block using ropivacaine preoperatively and postoperatively
  Arms: Group A
Drug: Morphine — Morphine intraoperatively and postoperatively
  Arms: Group B

SUMMARY:
60 patients ASA I-III, undergoing open nephrectomy will be randomly assigned into one of two groups, namely group A (n=30), where a thoracic paravertebral block will be performed preoperatively and a paravertebral catheter for continuous and patient controlled bolus local anesthetic (ropivacaine) doses will be inserted and group B (n=30) where morphine IV will be administered at the beginning and the end of operation and postoperatively through patient controlled IV doses. NRS scores in static and dynamic conditions, complications, patient satisfaction, oxidative stress (through lactic acid, superoxide dismutase, malondialdehyde) and NGAL pre- and postoperatively, will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Physical status according to American Society of Anesthesiologists (ASA) I-III
* Patients scheduled for open nephrectomy

Exclusion Criteria:

* Previous operation on same kidney
* Contraindication of paravertebral block or any of the agents used in the protocol
* BMI above 32
* Any concurrent malignancy not cured
* Serious psychiatric, mental and cognitive disorders
* Block failure
* Chronic pain
* Severe kidney disfunction

Ages: 14 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-03-09 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
Postoperative pain | 48 hours
  Numerical Rating Scale (NRS) scores (Range 0-10, 0=no pain, 10=the worse pain ever)
Oxidative stress - lactic acid (mmol/L) | 24 hours
Oxidative stress - superoxide dismutase (units/ml) | 24 hours
Oxidative stress - malondialdehyde (nmol/mg protein) | 24 hours
Oxidative stress - neutrophil gelatinase-associated lipocalin (NGAL) (ng/ml) | 24 hours

SECONDARY OUTCOMES:
Complications | 48 hours
Patient satisfaction | 48 hours
  Patients asked whether they would choose the same anaesthetic management in a future operation: Yes/No
Patient mobilization | 7 days
  Patient reporting time of first standing to the side of the bed
Intestinal function | 7 days
  Time of first passing of rectal gas, reported by the patient
Chronic pain | 6 months
  Using of Graded Chronic Pain Scale (GCPS) Grade 0: No pain in prior 6 months Grade 1: Low Intensity - Low Disability Grade II: High Intensity Characteristic Pain Intensity - Low Disability Grade III: High Disability - Moderately Limiting Grade IV: High Disability - Severely Limiting

CONTACTS AND LOCATIONS:
Locations (1):
- Asklepieion Hospital of Voula, Athens, Greece

IPD SHARING:
Plan to Share IPD: No